CLINICAL TRIAL: NCT02281474
Title: Open Label Dose Escalation of Nilotinib in Cognitively Impaired Parkinson Disease Patients With Elevated Cerebrospinal Fluid and Blood α-Synuclein
Brief Title: Nilotinib in Cognitively Impaired Parkinson Disease Patients 001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2014-001
Record Dates: First submitted 2014-10-27; First posted 2014-11-03 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Parkinson's Disease; Parkinson's Disease Dementia; Diffuse Lewy Body Disease
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 150mg dosing (Active Comparator): This arm will take 150mg of Nilotinib by mouth daily for the 6 month drug period to establish a safe and efficacious dose.
  Interventions: Drug: Nilotinib
- 300mg dosing (Active Comparator): This arm will take 300mg of Nilotinib by mouth daily for the 6 month drug period to establish a safe and efficacious dose.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib
  Other Names: Tasigna

SUMMARY:
This pilot study will test Nilotinib's ability to alter the abnormal protein build up in Parkinson disease and Diffuse Lewey Body Disease patients . Patients will receive Nilotinib at different doses for 6 months. Patients will then be tested to see if there is change in three areas: 1) has the disease symptoms changed. 2) has levels of a specific misfolded protein changed in the fluid around their brain and spine. 3) Have inflammatory markers changed in the patient's blood and fluid around their brain and spine. If successful, this drug could be used to slow down or stop the progression of disorders that involve abnormal collection of misfolded proteins. However, the main purpose of this pilot study is to check for the safety of using this medication at this level.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 40 to 90 with Idiopathic Parkinson's Disease (Significant Sinemet response) on a stable medication drug regimen L-dopa and/or Dopamine agonist (at least 1 month before enrollment with no new medication change) and with moderate to severe cognitive impairment (MOCA ≤24).

Inclusions criteria:

1. Written informed consent
2. Capability and willingness to comply with the study related criteria
3. Patients between the age of 40-90 y
4. Diagnosis of PD according to the UK Brain Bank Diagnostic Criteria
5. Early PD subjects with MMSE between 23-30.
6. Hoehn and Yahr stage <2
7. Stable treatment (>4 weeks) with MAO-B inhibitor (Selegeline up to 10mg/d or rasagiline up to 1 mg/d) allowable
8. Patients not needing dopamine agonist or levodopa therapy presently or at least for the next 6 months
9. Idiopathic PD with NO genetic mutations (autosomal recessive or dominant)
10. Detectable levels of CSF for blood and CSF Alpha-Synuclein

Exclusion Criteria:

1. Patients with a known genetic form of PD that does not involve alpha-synuclein.
2. Unwillingness to undergo lumbar punctures
3. Immeasurable CSF α-synuclein.
4. Presence of dementia or severe cognitive impairment that would not permit the patient to give adequate feedback for potential side effects.
5. Unwilling to be in an off state for UPDRS assessment.
6. Pre-menopausal women
7. Patients with autosomal recessive (PARKIN, PINK1 or DJ1) or dominant mutations (LRRK2)
8. Patients with hypokalemia, hypomagnesaemia, or long QT syndrome.
9. Concomitant drugs known to prolong the QT interval
10. Strong CYP3A4 inhibitors
11. Any drugs or foods that may interact with Nilotinib as stated in the Package Insert (PI).
12. Medical history of liver and pancreatic diseases.
13. Clinical signs indicating syndromes other than idiopathic PD, including supranucelar gaze palsy, signs of frontal dementia, history of stroke, head injury or encephalitis, cerebellar sings, early severe autonomic involvement, Babinski's signs.
14. History of any cardiovascular disease, including hypertension, myocardial infraction or cardiac failure, angina, arrhythmia.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in α-synuclein and Tau concentrations in the CSF and serum of patients | 6 months
  Working Hypothesis: PD patients have been shown to have elevated levels of α-synuclein in their CSF. Nilotinib has been shown to reduce α-synuclein and Tau in the gastrointestinal tract and central nervous system in animal models, and similarly, we propose will show changes in CSF and serum α-synuclein concentrations in nilotinib treated PD patients.

SECONDARY OUTCOMES:
Determine nilotinib's efficacy by improvement in motor and non-motor symptoms | 6 months
  Working Hypothesis: By following strict safety guidelines, monitoring patients through physical examinations, self-examinations, laboratory and neurological examinations, nilotinib will be a safe drug to use in patients with PD and PD related patients.
  Determine if any clinical benefit is observed in this small, short, limited clinical trial.
  Working Hypothesis: In cell culture and animal models of PD, dopaminergic neurons have shown increased cell death with accumulating α-synuclein. Therefore, PD patients treated with nilotinib, which lowers α-synuclein and Tau in vivo and in vitro studies, will have improvement or stabilization of their motor UPDRS and cognition.
Safety and tolerability, as measured by number of Participants with Adverse Events | 6 months
  Working Hypothesis: By following strict safety guidelines, monitoring patients through physical examinations, self-examinations, laboratory and neurological examinations, nilotinib will be a safe drug to use in patients with PD and PD related patients.
  Determine if any clinical benefit is observed in this small, short, limited clinical trial.
  Working Hypothesis: In cell culture and animal models of PD, dopaminergic neurons have shown increased cell death with accumulating α-synuclein. Therefore, PD patients treated with nilotinib, which lowers α-synuclein and Tau in vivo and in vitro studies, will have improvement or stabilization of their motor UPDRS and cognition.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102